CLINICAL TRIAL: NCT01966965
Title: Phase 3 Efficacy and Safety Study for PIOLIN® Shampoo to Treat Pediculosis
Brief Title: Efficacy and Safety Study for PIOLIN® Shampoo
Acronym: ESPX
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Phytopharm Consulting Brazil (Network)
Collaborators: Laboratório Saúde Ltda - principal e único patrocinador (Unknown)
Responsible Party: Principal Investigator, Karla F. Deud Jose, CEO, Phytopharm Consulting Brazil
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ESPX2013
Record Dates: First submitted 2013-10-17; First posted 2013-10-22 (Estimated); Last update posted 2013-10-23 (Estimated); Status verified 2013-10

CONDITIONS: PEDICULOSIS
Keywords: PIOLIN®, PEDICULOSIS, EFFICACY, SAFETY, PHYTOMEDICINE,; ARRUDA, RUTA
MeSH Terms: conditions — Lice Infestations

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- PIOLIN® (Experimental): PIOLIN® SHAMPOO 5 DAYS CONTINUOUSLY STOP A WEEK AND APPLY AGAIN
  Interventions: Drug: PIOLIN®
- NEDAX (Active Comparator): FOLLOWING THE LEAFLET TREATMENT
  Interventions: Drug: NEDAX

INTERVENTIONS:
Drug: PIOLIN® — PIOLIN® SHAMPOO 5 DAYS CONTINUOUSLY STOP A WEEK AND APPLY AGAIN
  Other Names: RUTA GRAVEOLENS STANDARDIZED FLUID EXTRACT
  Arms: PIOLIN®
Drug: NEDAX — AS SPECIFIED AT THE LEAFLET
  Other Names: PERMETRIN
  Arms: NEDAX

SUMMARY:
This study aims to demonstrate the therapeutic efficacy and safety of Shampoo PIOLIN ® in the treatment of human pediculosis. Will be treated 212 patients aged 2-60 years with the infestation, along with the people in your family life. All will be submitted to the dosing regimen recommended in the package insert. 100% of the sample shall be subjected to clinical evaluation through comb, pre and post treatment and monitored after thirty days for evaluation of safety and possible adverse effects that may arise related to any of the components of the formula.

The efficacy study is active comparator, non-inferiority.

ELIGIBILITY:
Inclusion Criteria:

* Volunteers healthy female and male ;
* Children between 2 and 17 years ;
* Increased from 18 years;
* Availability of volunteer to maintain a stable weight during the study period (ranging from less than 2 kg) ;
* Displays lice infestation on clinical examination ;
* Voluntary participation ;
* Signing the consent form and / or Free and Informed Consent ;
* Willingness to comply with study procedures ;
* Complying that researchers can make use of all the information nameless , including publication and comply with the use and storage of all information confidential .

Exclusion Criteria:

* Use paint or other chemicals on the hair in the last four weeks that precede the study ;
* Concomitant Therapy ;
* Women who are pregnant or intend to become pregnant during the study ;
* Infants ;
* Volunteers not willing to sign and adhere to the Statement of Consent ;
* Known hypersensitivity to the product ;
* Participation in any other clinical study ;
* Any other condition that the investigator decides that might interfere with the results or involving a risk to the volunteer study

Ages: 2 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 212 (Estimated)
Dates: Start 2014-07; Primary Completion 2014-09 (Estimated); Study Completion 2014-10 (Estimated)

PRIMARY OUTCOMES:
EFFICACY | 17 DAYS
  AFTER 17 DAYS OF TREATMENT PATIENTS SHOULD HAVE NO INFESTATION - clinically

SECONDARY OUTCOMES:
SAFETY | 30 DAYS
  IN THE END OF 30 DAYS TREATMENT PATIENTS WILL BE EVALUATED WITH BLOOD/URINE ANALYSIS FOR CHECKING ANY CHANGE - biochemistry, lab exams

CONTACTS AND LOCATIONS:
Overall Officials: MONICA M MENDES, MD MSc, Principal Investigator — UCPEL-UNIVERSIDADE CATÓLICA DE PELOTAS; ACHILLES GENTILINI NETO, MD, Study Chair — INDEPENDENT
Locations (1):
- Ubs Fatima, Pelotas, Rio Grande do Sul, Brazil

REFERENCES:
- See also: Brazilian researchers and professors site — http://lattes.cnpq.br/8425815106310226